CLINICAL TRIAL: NCT00733148
Title: Randomised Trial to Investigate the Correlation Between the Interstitial and Arterial Blood Concentrations of Glucose During Subcutaneous Microdialysis Glucose Monitoring in Post Surgery Patients at the Intensive Care Unit.
Brief Title: Correlation Between the Interstitial and Arterial Glucose in Post Surgery Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Thomas R. Pieber, Medical University of Graz
Other Study IDs: CM1
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Intensive Care
Keywords: glucose, interstitial, intensive care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Routine Care
  Interventions: Drug: dosing of insulin
- 2: Insulin infusion based on model predictive algorithm (MPC)
  Interventions: Drug: dosing of insulin

INTERVENTIONS:
Drug: dosing of insulin — Dosing od insulin is calculated by a computer based algorithm
  Other Names: Model predictive control

SUMMARY:
The EU funded project CLINICIP (Closed Loop Insulin Infusion for Critically Ill Patients) aims to develop a low-risk monitoring and control device which allows maintaining metabolic control in intensive care units. A system will be developed comprising three subsystems: a body interface for the delivery of biofluids, biosensors for the determination of glucose concentration in these biofluids and an adaptive control algorithm that generates advice and thus represents a decision support system with respect to insulin infusion rate to establish glycaemic control in critically ill patients. Within a closed loop system, intensified insulin treatment will make use of the calculations leading to external regulation of glucose.

It is the aim of this study to evaluate the correlation between arterial blood glucose concentrations and interstitial fluid glucose concentrations in post surgery patients in the Intensive Care Unit (ICU). Interstitial fluid glucose concentrations are based on microdialysis in subcutaneous adipose tissue and calculated using the ionic reference technique.

DETAILED DESCRIPTION:
This trial includes a screening visit (V1) and a monitoring visit (V2) and follow-up assessment. Visit 1 will be performed before performance of surgery to obtain informed consent and to assess patient eligibility. At Visit 2 monitoring visit after surgery) arterial blood glucose values will be monitored and subcutaneous sampling of ISF with microdialysis for glucose determination will be performed. Visit 2 will last from admittance to the ICU for 48 hours. In a follow-up assessment, two weeks after the end of visit 2, further clinical relevant data for the two week period after visit 2 will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities.
* Planned surgery and post-surgery stay in the ICU.
* Study day inclusion criteria: Increased blood glucose levels at admission to the ICU ( > 120 mg/dL; > 6.7 mM)
* Age of patients in the range from 18 to 90 years.

Exclusion Criteria:

* Known or suspected allergy against insulins.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
* Any disease or condition which the Investigator or the treating physician feels would interfere with the trial or the safety of the patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a blood glucose level of more than 120 mg/dl (6.7mM) at admission to the ICU after surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Time concentration profiles of arterial blood glucose concentrations and interstitial fluid glucose concentrations | hourly

SECONDARY OUTCOMES:
Prospectively calibrated interstitial fluid glucose concentration profiles | hourly

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Schaupp L, Plank J, Kohler G, Schaller R, Wrighton C, Ellmerer M, Pieber TR. Prediction of glucose concentration in post-cardiothoracic surgery patients using continuous glucose monitoring. Diabetes Technol Ther. 2011 Feb;13(2):127-34. doi: 10.1089/dia.2010.0117. PMID 21284479